CLINICAL TRIAL: NCT05214326
Title: A Real-World Study to Assess the Disease Control of Moderate to Severe Atopic Dermatitis in Patients Receiving Dupilumab Therapy, With Atopic Dermatitis Control Tool in Gulf Countries
Brief Title: A Study to Assess the Disease Control of Moderate to Severe Atopic Dermatitis in Male and Female Participants of Atleast 12 Years Old Receiving Dupilumab Injections in Gulf Countries
Acronym: AD-impaCT
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS17399; U1111-1269-6618 (Registry Identifier: ICTRP); OBS17399 (Other: Sanofi Identifier)
Record Dates: First submitted 2021-12-23; First posted 2022-01-28 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Dermatitis Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with moderate to severe atopic dermatitis: Participants initiating dupilumab therapy within 30 days of enrollment, according to the treating physician's decision independently of study participation.

SUMMARY:
Primary objective:

To assess the disease control of moderate to severe atopic dermatitis in patients aged 12 years and above treated with dupilumab therapy using Atopic Dermatitis Control Tool (ADCT) after 24 weeks of treatment.

Secondary objectives:

* To figure the proportion of patients with reduction of ADCT score by 5 points after 4, 12, and 24 weeks of treatment.
* To figure the proportion of patients with ADCT score less than 7 at weeks 4, 12, and 24.
* Assess the effectiveness of dupilumab in moderate to severe atopic dermatitis (AD) patients, using the severity score as routine practice SCORing Atopic Dermatitis (SCORAD).
* To describe comorbidities related to type 2 inflammation.
* To characterize the safety profile of dupilumab in the local Gulf population.
* To evaluate treatment satisfaction in the local Gulf population.

DETAILED DESCRIPTION:
24 weeks

ELIGIBILITY:
Inclusion Criteria:

* Having moderate to severe atopic dermatitis:

  * Moderate atopic dermatitis is defined at screening and baseline as i) Atopic dermatitis body surface area (BSA) involvement ≥10%; and ii) Pruritus numerical rating scale (NRS) ≥3, Eczema Area and Severity Index (EASI) score ≥16 at screening and baseline, Investigator's Global Assessment (IGA)=3, or SCORing Atopic Dermatitis (SCORAD) is between 25 and 50.
  * Severe atopic dermatitis is defined at screening and baseline as i) Atopic dermatitis BSA involvement ≥10%; ii) Eczema Area and Severity Index (EASI) score ≥20; iii) Investigator's Global Assessment (IGA) score = 4, or SCORAD ≥50.
* Initiating dupilumab therapy within 30 days of enrollment, according to the treating physician's decision independently of study participation.
* Participants and/or his legally approved representatives (LAR, in case of minor subject) agrees to sign an informed consent or an assent.
* Age of 12 years or above.

Exclusion Criteria:

* Participation in another trial.
* Pregnancy or lactating or planning/intending to be pregnant in the next 6 months.
* Presence of active chronic or acute infection requiring systemic treatment
* Diagnosed active endoparasites infection, or suspected high risk of infection.
* Human immunodeficiency virus (HIV), hepatitis B or C, malignancy, or other concomitant illnesses.

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with moderate to severe atopic dermatitis, initiating dupilumab therapy within 30 days of enrollment, according to the treating physician's decision independently of study participation.
Sampling Method: Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Percentage of patients achieving an Atopic Dermatitis Control Tool (ADCT) score less than 7 (defined as in control according to ADCT) | At week 24
  ADCT is a questionnaire to assess patient-self-perceived control of their atopic dermatitis (AD) with a total score from 0 to 24; higher scores indicate lower AD control.

SECONDARY OUTCOMES:
Percentages (%) of patients achieving a reduction of 5 points from baseline in ADCT | At weeks 4, 12, and 24
  ADCT is a questionnaire to assess patient-self-perceived control of their AD with a total score from 0 to 24; higher scores indicate lower AD control.
Percentages (%) of patients with ADCT score less than 7 | At weeks 4 and 12
  ADCT is a questionnaire to assess patient-self-perceived control of their AD with a total score from 0 to 24; higher scores indicate lower AD control.
Percentages (%) for patients achieving 50% and 75% reduction from baseline in SCORAD score (SCORAD-50 and SCORAD-75) | At week 24
  SCORAD is used to assess the extent and severity of AD. Extent and severity of AD as well as subjective assessment of symptoms were assessed and scored. SCORAD total score ranges from 0 (absent disease) to 103 (severe disease).
Mean change in SCORAD | From baseline (week 0) to week 24
  SCORAD is used to assess the extent and severity of AD. Extent and severity of AD as well as subjective assessment of symptoms were assessed and scored. SCORAD total score ranges from 0 (absent disease) to 103 (severe disease).
Number of patients with at least one type-2 inflammation comorbidity | Baseline (week 0) to week 24
  Comorbidities related to type-2 inflammation as (allergic rhinitis, bronchial asthma, chronic rhinosinusitis with nasal polyps, and eosinophilic esophagitis).
Adverse events (AEs) related to dupilumab use | Baseline (week 0) to week 24
  Number of patients experiencing adverse events (AEs) related to dupilumab use.
Serious adverse events (SAEs) related to dupilumab use | Baseline (week 0) to week 24
  Number of patients experiencing serious adverse events (SAEs) related to dupilumab use.
Adverse events of special interest (AESI) related to dupilumab use | Baseline (week 0) to week 24
  Number of patients experiencing adverse events of special interest (AESI) related to dupilumab use. An AESI is an adverse event (serious or non-serious) of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and rapid communication by the Investigator to the Sponsor is required.
Treatment interruption due to any adverse drug reaction (ADR), AE, SAE, or AESI | Baseline (week 0) to week 24
  Number of patients experiencing treatment interruption due to any adverse drug reaction, AE, SAE, or AESI. An AESI is an adverse event (serious or non-serious) of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and rapid communication by the Investigator to the Sponsor is required.
Treatment satisfaction: Number of patients achieving patient global assessment of treatment effect (PGATE) level very good | At week 24
  PGATE is an assessment tool used to rate the treatment effect of the medication on atopic dermatitis (AD), with scores ranging from 0 to 4 (0 = poor; 1 = fair; 2 = good; 3 = very good; 4 = excellent), i.e., higher score indicated higher treatment effect.

CONTACTS AND LOCATIONS:
Overall Officials: Trial Transparency Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- Investigational site Kuwait, Kuwait City, Kuwait
- Investigational site Saudi Arabia, Saudi Arabia, Saudi Arabia
- Investigational site United Arab Emirates, United Arab Emirates, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org